CLINICAL TRIAL: NCT05565768
Title: A Phase 1 Randomized, Placebo-Controlled Single Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of HZN-457 in Healthy Volunteers
Brief Title: Study to Evaluate HZN-457 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Horizon Therapeutics Ireland DAC (Industry)
Responsible Party: Sponsor
Organization: Horizon Pharma Ireland, Ltd., Dublin Ireland (Industry)
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Other
Other Study IDs: HZNP-HZN-457-101
Record Dates: First submitted 2022-09-26; First posted 2022-10-04 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HZN-457 (Experimental)
  Interventions: Drug: HZN-457
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HZN-457 — HZN-457 will be given in one subcutaneous administration
  Arms: HZN-457
Drug: Placebo — Placebo will be given in one subcutaneous administration
  Arms: Placebo

SUMMARY:
The purpose of this first in human study is to assess safety, pharmacokinetics, pharmacodynamics, and immunogenicity of single ascending doses of HZN-457.

ELIGIBILITY:
Inclusion Criteria:

* Screening serum uric acid (sUA) ≥ 4 mg/dL (238 µmol/L)
* Screening body mass index (BMI) between 20 to 34.0 kg/m2, inclusive
* Medically healthy with no clinically significant medical history, physical examination, laboratory profiles, vital signs, or ECG findings, as deemed by the Investigator.
* Male participants must refrain from donating sperm and either agree to remain abstinent from heterosexual intercourse OR agree to utilize contraception
* Female participants must be non-pregnant, non-lactating postmenopausal woman of non-childbearing potential (WONCBP) with a follicle-stimulating hormone (FSH) level in the postmenopausal range (> 40 IU/L)

Exclusion Criteria:

* History or presence of gout.
* Use of any prescription medication within 14 days or 5 half-lives prior to dosing
* Participation in another investigational clinical study (eg, drug, vaccine, invasive device) within 30 days or 5 half-lives, whichever is longer, prior to Day 1.
* Current liver disease, as determined by alanine transaminase (ALT) or aspartate transaminase (AST) levels > upper limit of normal (ULN) at Screening or Day -1.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2022-11-22 (Actual); Primary Completion 2023-08-09 (Actual); Study Completion 2023-08-09 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) and adverse events of special interest (AESIs) (injection site reactions (ISRs). | Day 1 up to Day 337
Change from Baseline in Hemoglobin value. | Baseline, Day 2, Day 4, Day 8, Day 15, Day 43, Day 85
Change from Baseline in white blood cell counts. | Baseline, Day 2, Day 4, Day 8, Day 15, Day 43, Day 85
Change from Baseline in platelet counts. | Baseline, Day 2, Day 4, Day 8, Day 15, Day 43, Day 85
Change from Baseline in Prothrombin Time. | Baseline, Day 2, Day 4, Day 8, Day 15, Day 43, Day 85
Change from Baseline in Activated Partial Thromboplastin Time. | Baseline, Day 2, Day 4, Day 8, Day 15, Day 43, Day 85
Change from Baseline in Aspartate Aminotransferase (AST) value. | Baseline, Day 2, Day 4, Day 8, Day 15, Day 43, Day 85
Change from Baseline in Alanine Aminotransferase (ALT) value. | Baseline, Day 2, Day 4, Day 8, Day 15, Day 43, Day 85
Change from Baseline in Urinalysis values. | Baseline, Day 2, Day 4, Day 8, Day 15, Day 43, Day 85
Change from Baseline in Systolic Blood Pressure values. | Baseline, Day 2, Day 4, Day 8, Day 15, Day 43, Day 85
Change from Baseline in Diastolic Blood Pressure values. | Baseline, Day 2, Day 4, Day 8, Day 15, Day 43, Day 85
Change from Baseline in Pulse Rate values. | Baseline, Day 2, Day 4, Day 8, Day 15, Day 43, Day 85
Change from Baseline in Respiratory Rate values. | Baseline, Day 2, Day 4, Day 8, Day 15, Day 43, Day 85
Change from Baseline in Body Temperature values. | Baseline, Day 2, Day 4, Day 8, Day 15, Day 43, Day 85
Change from Baseline in ECG Heart Rate values. | Baseline, Day 1 Post-Dose, Day 2, Day 4
Change from Baseline in ECG PR values. | Baseline, Day 1 Post-Dose, Day 2, Day 4
Change from Baseline in ECG QRS values. | Baseline, Day 1 Post-Dose, Day 2, Day 4
Change from Baseline in ECG QT values. | Baseline, Day 1 Post-Dose, Day 2, Day 4
Change from Baseline in ECG QTc values. | Baseline, Day 1 Post-Dose, Day 2, Day 4

SECONDARY OUTCOMES:
Peak plasma concentration (Cmax) | Day 1 to Day 8
Time to peak plasma concentration (Tmax) | Day 1 to Day 8
Area under the concentration-time curve from time 0 extrapolated to infinity (AUCinf) | Day 1 to Day 8
Elimination half-life (t1/2) | Day 1 to Day 8
Fraction of the administered dose excreted into the urine (Fe) | Day 1 to Day 2
Change and percent change from baseline in serum uric acid (sUA) evaluated post dosing | Day 1 to Day 337

CONTACTS AND LOCATIONS:
Overall Officials: Horizon Medical Director, Study Director — Horizon Therapeutics
Locations (2):
- New Zealand (2):
  - New Zealand Clinical Research, Auckland
  - New Zealand Clinical Research, Christchurch

IPD SHARING:
Plan to Share IPD: Undecided